CLINICAL TRIAL: NCT05819892
Title: Phase I Trial Testing the Safety and Tolerability of Chemoradiation Followed by Chemotherapy + Dostarlimab for Stage IIIC, Node Positive, Endometrial Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0618; NCI-2023-03071 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel; Carboplatin; dostarlimab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Adjuvant Therapy During Radiation (Experimental): Participants will receive an active treatment for 6 cycles. Participants will be on maintenance for 14 cycles, as long as the disease does not get worse. Follow-up will then occur every 6 months for 5 years (from your enrollment date).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Dostarlimab; Drug: Cisplatin
- Adjuvant Therapy After Radiation (Experimental): Participants will receive an active treatment for 6 cycles. Participants will be on maintenance for 14 cycles, as long as the disease does not get worse. Follow-up will then occur every 6 months for 5 years (from your enrollment date).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Dostarlimab; Drug: Cisplatin
- Immunotherapy after Radiation and Chemo (Experimental): Participants will receive an active treatment for 6 cycles. Participants will be on maintenance for 14 cycles, as long as the disease does not get worse. Follow-up will then occur every 6 months for 5 years (from your enrollment date).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Dostarlimab; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Given by IV (vein)
  Other Names: Taxol
Drug: Carboplatin — Given by IV (vein)
  Other Names: Paraplatin®
Drug: Dostarlimab — Given by IV (vein)
Drug: Cisplatin — Given by IV (vein)
  Other Names: Platinol®-AQ; Platinol®; CDDP

SUMMARY:
To learn if chemotherapy given in combination with radiation therapy, followed by maintenance therapy, can help to control endometrial cancer. The safety and effects of this study treatment will also be studied

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of this study is to describe the safety and toxicity of chemoradiation with concurrent immunotherapy, followed by chemotherapy plus concurrent immunotherapy, followed by immunotherapy maintenence in patients with stage IIIC endometrial cancer.

Secondary Objectives:

The secondary objectives are listed below.

* To estimate progression free survival
* To describe the time to recurence and the recurrence patterns including extent and location (i.e. isolated versus multi-focal, pelvic versus distant)
* To estimate disease specific survival and overall survival

Exploratory:

* To determine if the presence of deficient mismatch repair (dMMR) or microsatellite instability correlates with progression free survival, disease free survival and 5-year overall survival
* To assess patient reported outcomes (PROs) during the course of treatment and follow up

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to participate on this study only if they meet all of the following inclusion criteria.

1. Has read and understands the informed consent form (ICF) and has given written informed consent prior to any study procedures
2. Have surgically staged IIIC, pathologically confirmed endometrial cancer of any histologic subtype and be eligible for adjuvant chemoradiation followed by chemotherapy (Note: Surgical staging is defined as total hysterectomy and lymph node assessment.)
3. Enrolled within 8 weeks of surgery and started treatment within 10 weeks of surgery
4. Age ≥ 18 years
5. Performance Status of ECOG 0 or 1 (see Performance Status Criteria)
6. Adequate hematologic function within 14 days prior to enrollment defined as follows:

   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥ 100,000/mcl
   * Absolute neutrophil count (ANC) ≥ 1,500/mcl
7. Adequate renal function within 14 days prior to enrollment defined as follows: Creatinine

   ≤ 2 x laboratory upper limit of normal (ULN) or CrCl ≥60ml/min
8. Adequate hepatic function within 14 days prior to enrollment defined as follows:

   * Bilirubin ≤ 1.5 x ULN (patients with known Gilbert's disease who have bilirubin level ≤ 2 x ULN may be enrolled)
   * ALT and AST ≤ 2.5 x ULN
9. Adequate coagulation within 14 days prior to enrollment defined as INR or PT/aPTT ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
10. Prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial (i.e. non-melanomatous skin cancer).

Exclusion Criteria:

Patients are not eligible to participate on this study if they meet any of the following exclusion criteria.

1. Has not recovered (i.e., to Grade ≤ 1 or to baseline) from prior radiation, major surgery and chemotherapy-induced AEs.
2. Surgery ≤ 3 weeks prior to initiating protocol therapy Investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to initiating protocol therapy.
3. Has received prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapeutic antibody or other similar agents.
4. Has a history of a severe hypersensitivity reaction to monoclonal antibody or dostarlimab and/or its excipients.
5. Have active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. This includes, but is not limited to: a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, GuillainBarre syndrome, myasthenia gravis, systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome because of the risk of recurrence or exacerbation of disease.
6. History of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies.
7. Have a diagnosis of immunodeficiency or are receiving daily systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment:

   * Steroids received as CT scan contrast premedication may be enrolled.
   * The use of inhaled or topical corticosteroids is allowed.
   * The use of mineralocorticoids (e.g., fludrocortisone) for orthostatic hypotension or adrenocortical insufficiency is allowed.
   * The use of physiologic doses of corticosteroids may be allowed and in consultation with the study chair (e.g. 10 mg of prednisone used for replacement therapy for adrenal insufficiency).
8. Have received a live vaccine within 30 days of starting trial therapy.
9. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; and cirrhosis.

   --Evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load, tested positive for the presence of hepatitis B surface antigen, or have a positive hepatitis C antibody test result at screening or within 3 months prior to the first dose of study treatment.
10. Uncontrolled intercurrent illness including (but not limited to): ongoing or active infection (except for uncomplicated urinary tract infection), interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Have received any of the prohibited medications listed in Section 7.2.
12. Has leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiologic signs of CNS hemorrhage. Note: Asymptomatic brain metastases (i.e, off corticosteroids and anticonvulsants for at least 7 days) are permitted.
13. Known human immunodeficiency virus (HIV)-infected patients.
14. Women of childbearing potential (WoCBP) who have been not been permanently or surgically sterilized and are capable of procreation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Soliman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org